CLINICAL TRIAL: NCT01691690
Title: Analgesic Effect of Single Dose Intravenous Acetaminophen in Pediatric Patients Undergoing Tonsillectomy
Brief Title: Analgesic Effect of IV Acetaminophen in Tonsillectomies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Arlyne Thung, Clinical Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB12-00097
Record Dates: First submitted 2012-05-30; First posted 2012-09-25 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Adenotonsillitis; Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Acetaminophen; Midazolam; Sevoflurane; Nitrous Oxide; Oxygen; Propofol; Morphine; Ondansetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): Patients will receive pre-medication with oral midazolam Participants of this experimental arm of the study will receive Acetaminophen IV to evaluate opioid-sparing effect and pain score reduction..
  Interventions: Drug: Acetaminophen (paracetamol); Drug: Midazolam; Drug: Sevoflurane; Drug: Nitrous Oxide/Oxygen; Drug: Propofol; Drug: Morphine; Drug: Ondansetron; Drug: Dexamethasone
- Saline placebo infused intraoperatively (Placebo Comparator): For this arm Morphine will be administered to manage pain.
  Interventions: Drug: Normal Saline Flush; Drug: Midazolam; Drug: Sevoflurane; Drug: Nitrous Oxide/Oxygen; Drug: Propofol; Drug: Morphine; Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Acetaminophen (paracetamol) — Acetaminophen IV (15 mg/kg).
  Arms: IV Acetaminophen
Drug: Normal Saline Flush — Saline placebo will be infused intraoperatively.
  Arms: Saline placebo infused intraoperatively
Drug: Midazolam — Midazolam (0.5mg/kg to maximum dose of 20mg) given 15-20 minutes before induction.
  Other Names: Versed
Drug: Sevoflurane — Sevoflurane for anesthesia induction.
Drug: Nitrous Oxide/Oxygen — Combination of NO2 & O2 for anesthesia induction.
Drug: Propofol — Propofol 1-1.5 mg/kg to facilitate endotracheal intubation.
Drug: Morphine — Morphine 0.1 mg/kg given prior to intubation.
Drug: Ondansetron — Ondansetron (0.15 mg/kg, maximum dose of 4 mg) for postoperative nausea prophylaxis.
  Other Names: Zofran
Drug: Dexamethasone — Dexamethasone (0.25 mg/kg, maximum dose of 20 mg) for postoperative nausea prophylaxis.

SUMMARY:
Acetaminophen (paracetamol) is a first-line antipyretic and analgesic for mild and moderate pain for pediatric patients. Its common use (particularly in oral form) is underscored by its wide therapeutic window, safety profile, over the counter accessibility, lack of adverse systemic effects (as compared with NSAIDS and opioids) when given in appropriate doses.

Although the exact anti-nociceptive mechanisms of acetaminophen continue to be elucidated, these mechanisms appear to be multi-factorial and include central inhibition of the cyclo-oxygenase (COX) enzyme leading to decreased production of prostaglandins from arachidonic acid, interference with serotonergic descending pain pathways, indirect activation of cannabinoid 1 (CB1) receptors and inhibition of nitric oxide pathways through N-methyl-D-aspartate (NMDA) or substance P. Of the above mechanisms, the most commonly known is that of central inhibition of COX enzymes by which the decreased production of prostaglandins diminish the release of excitatory transmitters of substance P and glutamate which are both involved in nociceptive transmission (Anderson, 2008; Smith, 2011).

To date, several studies have shown acetaminophen's opioid sparing effect in the pediatric population when given by the rectal or intravenous routes (Korpela et al, 1999; Dashti et al, 2009; Hong et al, 2010).

DETAILED DESCRIPTION:
Once enrolled, subjects will have a standardized anesthetic on the day of surgery:

1. Pre-medication with oral midazolam (0.5mg/kg to maximum dose of 20mg) given 15-20 minutes before induction
2. Inhalation induction with sevoflurane and a mixture of N20/02
3. Propofol 1-1.5 mg/kg to facilitate endotracheal intubation
4. Morphine 0.1 mg/kg given prior to intubation
5. Maintenance anesthesia with isoflurane, titrated to 0.8-1 Minimal Anesthetic Concentration (MAC) with a mixture of Air/02
6. Acetaminophen IV (15 mg/kg) vs. saline placebo infused intraoperatively (randomized by pharmacy)
7. Ondansetron (0.15 mg/kg, maximum dose of 4 mg) and dexamethasone (0.25 mg/kg, maximum dose of 20 mg) for postoperative nausea prophylaxis.

Following surgery and extubation, baseline vitals will be obtained and pain scores will be assessed in the post anesthesia care unit (PACU) via Faces, Legs, Activity, Cry, Consolability Scale (FLACC).The presence of emergence delirium will be assessed via Pediatric Agitation and Emergence Delirium scale (PAED). Those subjects whose pain score is assessed at < 4 will receive standard postoperative care and no analgesics. Assessed pain scores > 4 will receive 0.5mcg/kg fentanyl q10 minutes as needed. Variables such as time to extubation in the PACU, time to first analgesic delivery, pain scores, # times/total dose of opioids given, presence of sedation, nausea/vomiting, duration of oxygen requirement in PACU, whether or not patient was discharged to floor on oxygen and total PACU time will be recorded during the duration of the patient's PACU stay. Subjects will be discharged to the inpatient floor from the PACU once standard discharge criteria have been met.

Following discharge from the PACU, standardized analgesics will be given for breakthrough pain (oral oxycodone 0.1mg/kg q4hrs pro re nata (PRN) pain). Enrolled patients will be followed during the duration of their inpatient stay. Duration of oxygen requirement on the floor, pain scores and number of administered oxycodone doses on the floor will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 2 years and younger than 9 years old requiring postoperative admission for tonsillectomy or adenotonsillectomy.
2. Functional status as assigned by the American Society of Anesthesiology (ASA) classification of I (1), II (2) or III (3).
3. Have a parent/guardian who are able to provide written informed consent in accordance with Human Investigations Committee/Institutional Review Board (HIC/IRB) regulations.
4. Have parent/guardian who are compliant with routine medical care, capable of subjective evaluation and able to read, understand and sign the informed consent.

Exclusion Criteria:

1. Male or female patients age greater than 9 years.
2. Have an American Society of Anesthesiologists Physical Status > IV (4)(severe disease that is life threatening).
3. Have a known hypersensitivity or allergy to acetaminophen.
4. Have a known allergy or intolerance to morphine or fentanyl.
5. Have received chronic opioid analgesic therapy prior to surgery.
6. Have renal disease.
7. Have hepatic disease.
8. Are morbidly obese (% BMI > 95).

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlyne Thung, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Anderson BJ. Paracetamol (Acetaminophen): mechanisms of action. Paediatr Anaesth. 2008 Oct;18(10):915-21. doi: 10.1111/j.1460-9592.2008.02764.x. PMID 18811827
- [Background] Smith HS. Perioperative intravenous acetaminophen and NSAIDs. Pain Med. 2011 Jun;12(6):961-81. doi: 10.1111/j.1526-4637.2011.01141.x. Epub 2011 May 31. PMID 21627768
- [Background] Korpela R, Korvenoja P, Meretoja OA. Morphine-sparing effect of acetaminophen in pediatric day-case surgery. Anesthesiology. 1999 Aug;91(2):442-7. doi: 10.1097/00000542-199908000-00019. PMID 10443608
- [Background] Dashti GA, Amini S, Zanguee E. The prophylactic effect of rectal acetaminophen on postoperative pain and opioid requirements after adenotonsillectomy in children. Middle East J Anaesthesiol. 2009 Jun;20(2):245-9. PMID 19583073
- [Background] Hong JY, Kim WO, Koo BN, Cho JS, Suk EH, Kil HK. Fentanyl-sparing effect of acetaminophen as a mixture of fentanyl in intravenous parent-/nurse-controlled analgesia after pediatric ureteroneocystostomy. Anesthesiology. 2010 Sep;113(3):672-7. doi: 10.1097/ALN.0b013e3181e2c34b. PMID 20693884

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Acetaminophen: Patients will receive pre-medication with oral midazolam. Participants of this experimental arm of the study will receive Acetaminophen IV to evaluate opioid-sparing effect and pain score reduction.
  Acetaminophen (paracetamol): Acetaminophen IV (15 mg/kg) will be infused intraoperatively over 15 minutes to evaluate the opioid-sparing effect and pain score reduction in pediatric patients undergoing tonsillectomy or adenotonsillectomy procedures.
  Morphine (hydromorphone): Morphine (0.1 mg/kg) will be added to manage pain prior to intubation.
- Saline Placebo: Patients will receive pre-medication with oral midazolam. Participants of this control arm will receive saline to establish a control model for evaluating opioid-sparing effect and pain score reduction compared to the intervention arm.
  Sodium Chloride (saline): 0.9% Sodium Chloride Placebo will be infused intraoperatively over 15 minutes to establish a control model while evaluating the pain score differences in pediatric patients undergoing tonsillectomy or adenotonsillectomy procedures.
  Morphine (hydromorphone): Morphine (0.1 mg/kg) will be added to manage pain prior to intubation.
Period: Overall Study
Arm/Group | IV Acetaminophen | Saline Placebo
Started | 125 | 125
Completed | 118 | 121
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Saline Placebo | Total
Number analyzed (Participants) | 118 | 121 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.87 (1.53) | 4.84 (1.42) | 4.855 (1.476)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 56 | 62 | 118
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 109.31 (10.82) | 108.78 (10.37) | 109.04 (10.58)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 18.85 (4.74) | 18.27 (4.02) | 18.56 (4.39)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: Kg/m2] | 15.56 (1.58) | 15.29 (1.36) | 15.42 (1.47)
Procedure time (min) [Mean (Standard Deviation); unit: minutes] | 15.85 (5.78) | 16.65 (5.90) | 16.26 (5.85)
Extubation time (min) [Mean (Standard Deviation); unit: minutes] | 16.65 (7.68) | 15.38 (8.52) | 16.01 (8.12)
Post-Anesthetic Care Unit time (min) [Mean (Standard Deviation); unit: minutes] | 64.57 (23.41) | 65.07 (19.40) | 64.82 (21.44)
Time to first analgesic on unit (min) [Mean (Standard Deviation); unit: minutes] | 298.36 (97.52) | 297.09 (106.91) | 297.74 (101.97)

OUTCOME MEASURES:

1. Primary Outcome: FLACC Pain Score Greater Than or Equal to 4
Description: The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. 5 pain measurements were performed at 0, 5, 15, 30, and 60 minutes after PACU arrival. This is the number of participants who reached a FLACC score >/= 4 at one or more time points.
Time Frame: 0-60 mins post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Saline Placebo
Number analyzed (Participants) | 118 | 121
Participants | 58 | 69

2. Secondary Outcome: Analgesics Administered After Arrival to Inpatient Ward and Number of Participants Requiring Each
Description: Analgesics administered after arrival to the inpatient ward included hydrocodone/acetaminophen, oxycodone, NSAIDS, acetaminophen, and morphine.
Time Frame: 8-12 hours post-operatively
Population: Comparing both groups for the time study subjects required breakthrough pain medication on the ward.
Measure: Count of Participants; unit: Participants
Groups:
- Saline Placebo Infused Intraoperatively: Patients will receive pre-medication with oral midazolam. Participants of this control arm will receive saline to establish a control model for evaluating opioid-sparing effect and pain score reduction compared to the intervention arm.
  Sodium Chloride (saline): 0.9% Sodium Chloride Placebo will be infused intraoperatively over 15 minutes to establish a control model while evaluating the pain score differences in pediatric patients undergoing tonsillectomy or adenotonsillectomy procedures.
  Morphine (hydromorphone): Morphine (0.1 mg/kg) will be added to manage pain prior to intubation.
Arm/Group | IV Acetaminophen | Saline Placebo Infused Intraoperatively
Number analyzed (Participants) | 118 | 120
Participants
  hydrocodone/acetaminophen | 68 | 57
  oxycodone | 31 | 39
  NSAIDS | 15 | 22
  acetaminophen | 3 | 2
  morphine | 1 | 0

3. Secondary Outcome: Time of First Opioid Analgesia in PACU
Description: Mean time to first drug administration among patients requiring opioid analgesia in the PACU.
Time Frame: 0-90 minutes post-operatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IV Acetaminophen | Saline Placebo Infused Intraoperatively
Number analyzed (Participants) | 118 | 121
minutes | 56.80 (14.15) | 60.46 (20.51)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each patient from pre-operative registration, peri-operatively, until hospital discharge post-operatively (Data collection occurred over the course of a 24 hour period).
Arm/Group | IV Acetaminophen | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/121
Other Adverse Events (participants affected / at risk) | 11/118 | 16/121
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen (N=118) | Saline Placebo (N=121)
Post-operative nausea or vomiting (PONV) (General disorders) | 1 | 4
Respiratory complications (Respiratory, thoracic and mediastinal disorders) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No